CLINICAL TRIAL: NCT02961829
Title: Multi Interventional Study Exploring HIV-1 Residual Replication: a Step Towards HIV-1 Eradication and Sterilizing Cure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Ricardo Sobhie Diaz, MD, PHD, Associate Professor of Medicine, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPARC-7
Record Dates: First submitted 2015-12-18; First posted 2016-11-11 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Chronic Infection; HIV
Keywords: Dendritic Cell vaccination using; antiretroviral intensification; Auranofin; Histone Deacetylase Inhibitor; residual viral replication; HIV sanctuaries; HIV latency
MeSH Terms: conditions — Persistent Infection | interventions — Maraviroc; dolutegravir; lentiviral minigene vaccine of COVID-19 coronavirus; Auranofin; Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Antiretroviral Treated (ART) Group (No Intervention): Five patients will receive no further intervention this group (control group)
- ART Intensification Group (Experimental): Five patients will receive antiretroviral intensification with maraviroc and dolutegravir for 48 weeks
  Interventions: Drug: Maraviroc; Drug: Dolutegravir
- ART Intensification + Nicotinamide Group (Experimental): Five patients will receive antiretroviral intensification with maraviroc and dolutegravir and the Sirtuin Histone deacetylase inhibitor nicotinamide for 48 weeks.
  Interventions: Drug: Maraviroc; Drug: Dolutegravir; Drug: Sirtuin Histone deacetylase inhibitor
- ART Intensification + Auranofin Group (Experimental): Five patients will receive antiretroviral intensification with maraviroc and dolutegravir for 48 weeks and the gold salt auranofin for 24 weeks.
  Interventions: Drug: Maraviroc; Drug: Dolutegravir; Drug: Auranofin
- ART Intensification + DC vaccine Group (Experimental): Five patients will receive antiretroviral intensification with dolutegravir and for 48 weeks, and dendritic cell vaccine.
  Interventions: Drug: Dolutegravir; Biological: Dendritic Cell Vaccine
- Multi Interventional Group (Experimental): Five patients will receive antiretroviral intensification with dolutegravir and the Sirtuin Histone deacetylase inhibitor nicotinamide for 48 weeks, and gold salt for 24 weeks and dendritic cell vaccine.
  Interventions: Drug: Dolutegravir; Biological: Dendritic Cell Vaccine; Drug: Auranofin; Drug: Sirtuin Histone deacetylase inhibitor

INTERVENTIONS:
Drug: Maraviroc — antiretroviral intensification
  Other Names: Selzentry; Celsentri
  Arms: ART Intensification + Auranofin Group; ART Intensification + Nicotinamide Group; ART Intensification Group
Drug: Dolutegravir — antiretroviral intensification
  Other Names: Tivicay
  Arms: ART Intensification + Auranofin Group; ART Intensification + DC vaccine Group; ART Intensification + Nicotinamide Group; ART Intensification Group; Multi Interventional Group
Biological: Dendritic Cell Vaccine — Therapeutic vaccination
  Other Names: DC Vaccine
  Arms: ART Intensification + DC vaccine Group; Multi Interventional Group
Drug: Auranofin — purging
  Other Names: Gold Salt
  Arms: ART Intensification + Auranofin Group; Multi Interventional Group
Drug: Sirtuin Histone deacetylase inhibitor — latency disruption
  Other Names: Nicotinamide
  Arms: ART Intensification + Nicotinamide Group; Multi Interventional Group

SUMMARY:
It is becoming clear that a combination of interventions will be desirable to achieve HIV cure. Therefore the investigators propose a pilot proof of concept study, using combination of a number of different interventions for eradicating residual plasma viremia and decreasing HIV reservoirs. The investigators hypothesize that, (i) antiretroviral intensification using Maraviroc, and/or dolutegravir with (ii) Dendritic Cell vaccination using autologous HIV, and (iii) purging intervention using the Class III HDACs, Sirtuin-1, and (iv) decreasing the ratio of long-lived central memory (TCM)/transitional memory (TTM) CD4+ T-cells using Auranofin will provide a synergistic impact leading to a sterilizing cure of HIV infection. Results of this study may provide insightful evidence for planning the next steps using the more efficacious combination of intervention strategies towards HIV sterilizing cure.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old Documented HIV-1 infection.
* Has voluntarily signed ICF.
* On HAART ≥ 2 years, without changes in the 24 weeks immediately prior to screening.
* HIV viral load <50 copies/mL, and never > 50 copies/mL on 2 consecutive occasions in the last 2 years. CD4 count nadir.
* > 350 cells/ mm3 Current CD4 count > 500 cells/ mm3.
* R5 HIV-1 at Screening as defined by proviral DNA genotropism.

Exclusion Criteria:

A subject will NOT be eligible for study participation if he/she meets ANY of the following criteria:

* Any evidence of an active AIDS-defining condition.
* Any significant acute medical illness in the past 8 weeks.
* Women who are pregnant or breastfeeding.
* Use of any of the following within 90 days prior to entry: systemic cytotoxic chemotherapy; investigational agents; immunomodulators (colony-stimulating factors, growth factors, systemic corticosteroids, HIV vaccines, immune globulin, interleukins, interferons); coumadin, warfarin, or other Coumadin derivative anticoagulants. Use of an agent definitely or possibly associated with effects on QT intervals: amiodarone, arsenic trioxide, astemizole, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide, dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, probucol, procainamide, quinidine, sotalol, sparfloxacin, terfenadine, thioridazine.
* Receipt of compounds with HDAC inhibitor-like activity, such as valproic acid or nicotinamide within the last 30 days. Potential participants may enroll after a 30-day washout period.
* Known hypersensitivity to the components of gold salt, nicotinamide or its analogs.
* Hepatitis B (HBsAg +) or Hepatitis C (HCV RNA +) infection.
* Known renal insufficiency defined as calculated creatinine clearance (Cockcroft Gault formula) <60 mL/min.
* Subjects with a laboratory abnormality grade 3 or 4 with the following exceptions: pancreatic amylase, cholesterol, triglyceride, gamma glutamyl transpeptidase, bilirubin.
* Any condition which, in the investigators opinion, could compromise the subject's safety or adherence to the trial protocol.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Ultrasensitive RNA Viral load, | from baseline and every 4 weeks up to 48 weeks.
Cell-associated HIV RNA | from baseline and every 4 weeks up to 48 weeks.
Episomal DNA | from baseline and every 4 weeks up to 48 weeks
specific HIV antibodies | from baseline and every 4 weeks up to 48 weeks
CD38 and HLA-DR on CD4 and CD8+ cells | from baseline and every 4 weeks up to 48 weeks
PBMC for env sequence evolution | from baseline and every 4 weeks up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CCDI, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Almeida Baptista MV, da Silva LT, Samer S, Oshiro TM, Shytaj IL, Giron LB, Pena NM, Cruz N, Gosuen GC, Ferreira PRA, Cunha-Neto E, Galinskas J, Dias D, Sucupira MCA, de Almeida-Neto C, Salomao R, da Silva Duarte AJ, Janini LM, Hunter JR, Savarino A, Juliano MA, Diaz RS. Immunogenicity of personalized dendritic-cell therapy in HIV-1 infected individuals under suppressive antiretroviral treatment: interim analysis from a phase II clinical trial. AIDS Res Ther. 2022 Jan 12;19(1):2. doi: 10.1186/s12981-021-00426-z. PMID 35022035
- [Derived] Diaz RS, Shytaj IL, Giron LB, Obermaier B, Della Libera E Jr, Galinskas J, Dias D, Hunter J, Janini M, Gosuen G, Ferreira PA, Sucupira MC, Maricato J, Fackler O, Lusic M, Savarino A; SPARC Working Group. Potential impact of the antirheumatic agent auranofin on proviral HIV-1 DNA in individuals under intensified antiretroviral therapy: Results from a randomised clinical trial. Int J Antimicrob Agents. 2019 Nov;54(5):592-600. doi: 10.1016/j.ijantimicag.2019.08.001. Epub 2019 Aug 5. PMID 31394172